CLINICAL TRIAL: NCT04941937
Title: Selinexor in Combination With Immunomodulator to Treat Relapsed/Refractory Multiple Myeloma Patients
Brief Title: Selinexor in Combination With Immunomodulator （Thalidomide/Pomalidomide/Lenalidomide）in RRMM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juan Du (Other)
Responsible Party: Sponsor-Investigator, Juan Du, Chief physician, professor, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-IIT-MM-004
Record Dates: First submitted 2021-06-25; First posted 2021-06-28 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
Keywords: Selinexor（ATG-010）; Multiple Myeloma; Relapsed/Refractory Multiple Myeloma; Thalidomide; Pomalidomide; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Thalidomide; Lenalidomide; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm I: Selinexor+Thalidomide+Dexamethasone (Experimental): Arm I is given XTd regimen Selinexor 60mg/d QW, Thalidomide 100mg/d, d1-28 and Dexamethasone 40mg/d QW) in approximately 30 subjects. 4 weeks per cycle and include a total of 12 cycles.
  Interventions: Drug: Selinexor; Drug: Thalidomide; Drug: Dexamethasone
- Arm II: Selinexor+Lenalidomide+Dexamethasone (Experimental): Arm II is given XRd regimen Selinexor 60mg/d QW, Lenalidomide 25mg/d, d1-21 and Dexamethasone 40mg/d QW) in approximately 30 subjects. 4 weeks per cycle and include a total of 12 cycles.
  Interventions: Drug: Selinexor; Drug: Lenalidomide; Drug: Dexamethasone
- Arm III: Selinexor+Pomalidomide+Dexamethasone (Experimental): Arm III is given XPd regimen Selinexor 60mg/d QW, Pomalidomide 4mg/d, d1-21 and Dexamethasone 40mg/d QW) in approximately 30 subjects. 4 weeks per cycle and include a total of 12 cycles.
  Interventions: Drug: Selinexor; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor (ATG-010# is a first-in-class, oral selective exportin 1 (XPO1) inhibitor (1,2). Selinexor functions by binding with and inhibiting the nuclear export protein XPO1 (also called CRM1), leading to the accumulation of tumor suppressor proteins in the cell nucleus along with inhibition of translation of oncoprotein mRNAs. Selinexor 60mg/d QW
  Other Names: ATG-010/KPT-330
Drug: Thalidomide — 100mg/d, Po. on day1-28
  Other Names: fǎn yìng tíng
  Arms: Arm I: Selinexor+Thalidomide+Dexamethasone
Drug: Lenalidomide — PO,Lenalidomide 25mg once daily from D1-21
  Other Names: Revlimid; An xian
  Arms: Arm II: Selinexor+Lenalidomide+Dexamethasone
Drug: Pomalidomide — Pomalidomide will be given at 4mg once daily for 21 days in a 28-day cycle, PO.
  Other Names: POMALYST
  Arms: Arm III: Selinexor+Pomalidomide+Dexamethasone
Drug: Dexamethasone — Dexamethasone will be given at a dose of 40mg orally once a week for 4 weeks (D1,8,15,22).
  Other Names: Dex

SUMMARY:
Multiple myeloma (MM) is an incurable plasma cell cancer that almost all patients eventually relapse despite advancement in treatment strategies. B-cell maturation antigen (BCMA) is a cell surface receptor that expressed primarily by malignant and normal plasma cells. This is a single-arm that includes three arms, Selinexor(ATG-010) in Combination with Immunomodulator (Thalidomide/ Pomalidomide/ Lenalidomide）and Dexamethasone to Treat Relapsed/Refractory Multiple Myeloma Patients. To evaluate efficacy and safety of Selinexor in combination with Immunomodulator and Dexamethasone in RRMM patients received at least one prior lines of therapy.

DETAILED DESCRIPTION:
This is a single-arm and open-label phase II study of Relapsed/Refractory Multiple Myeloma patients who have received at least one prior lines of treatment therapy; This study includes three experimental arms. Arm I is given XTd regimen (ATG-010 60mg/d QW, Thalidomide 100mg/d and Dexamethasone 40mg/d QW) in approximately 30 subjects. Arm II is given XRd regimen (ATG-010 60mg/d QW, Lenalidomide 25mg/d d1-21 and Dexamethasone 40mg/d QW) in approximately 30 subjects, Arm III is given XPd（ATG-010 60mg/d QW, Pomalidomide 4mg/d d1-21 and Dexamethasone 40mg/d QW ) in approximately 30 subjects,The three arms are 4 weeks per cycle and include a total of 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

  1. Known and written informed consent (ICF) voluntarily.
  2. Age ≥ 18 years and ≤ 75 years.
  3. Patients with multiple myeloma who have received first-line treatment (induction, autologous transplantation and maintenance as the same first-line treatment) and achieved at least partial remission in induction.
  4. At or after accepting first-line regimen, subjects must have progression disease (PD) recorded which is determined by researcher according to IMWG criteria.
  5. Any clinically significant non-hematological toxicities (except for hair loss, peripheral neuropathy, which is otherwise stipulated in Article 13 of the exclusion criteria) that relevant to previous therapies must have resolved to ≤Grade 2 prior to first dose of study drug.
  6. Left ventricular ejection fraction#LVEF #≥50% by an echocardiogram or MUGA scan in 42 days before the first administration
  7. Adequate hepatic function: total bilirubin < 2× upper limit of normal (ULN) (for patients with Gilbert's syndrome, a total bilirubin of < 3× ULN is required), AST < 2.5× ULN, and ALT < 2.5× ULN.
  8. Adequate renal function: estimated creatinine clearance ≥ 20 mL/min (calculated using the formula of Cockroft-Gault).
  9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
  10. Measurable MM as defined by at least one of the following:

      1. Serum M-protein (SPEP) ≥ 10 g/L
      2. 24 hours-Urinary M-protein excretion ≥ 0.2 g (200 mg)
      3. Serum FLC ≥ 100 mg/L with abnormal FLC ratio
  11. Expected survival is more than 6 months.
  12. Adequate hematopoietic function (no blood transfusion within 2 weeks and no G-CSF/GM-CSF supportive treatment within 1 week prior to screening test):

      1. Hemoglobin level ≥ 80 g/L
      2. ANC ≥ 1,000/mm3 (1.0×109/L)
      3. Platelet count ≥ 75,000/mm3 (75×109/L)
  13. Female patients of childbearing potential must meet below two criteria:

      1. must agree to use effective contraception methods since signature in ICF, throughout the study and for 3 months following the last dose of study treatment.
      2. must have a negative serum pregnancy test at screening. Note: A woman is considered of childbearing potential following menarche and until becoming postmenopausal (defined as no menstrual period for a minimum of 12 months) or permanently sterile (having undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy). A woman who is taking oral contraceptive or using intrauterine device is considered of childbearing potential.
  14. Male patients (including those who have received vasectomy) must use a condom if sexually active with a female of child-bearing potential throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

* Patients who meet any of the following criteria will not be enrolled:

  1. Asymptomatic (smoldering) MM.
  2. Plasma cell leukemia.
  3. Documented active amyloidosis.
  4. Previously refractory or intolerant to immunomodulators.
  5. Pregnancy or breastfeeding.
  6. Major surgery was performed within 4 weeks prior to the first study.
  7. Patients with active, unstable cardiovascular diseases, fits any of the following:

     1. Symptomatic ischemia, or
     2. Uncontrolled clinically-significant conduction abnormalities (e.g., patients with ventricular tachycardia on antiarrhythmics are excluded; patients with first-degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) are allowed), or
     3. Congestive heart failure (CHF) of New York Heart Association (NYHA) ≥ Grade 3, or
     4. Acute myocardial infarction (AMI) within 3 months prior to the first dose of study drug.
  8. Uncontrolled active infection within 1 week prior to the first dose of study drug.
  9. Known HIV positive.
  10. Known active hepatitis A, B, or C infection; or known positive for HCV RNA or HBsAg. (Note: patients with HBsAg negative but HBc Ab positive need further HBV-DNA test, excluded if HBV-DNA ≥103 , if HBV-DNA # 103 need anti-viral drugs)
  11. Prior malignancy that required treatment or has shown evidence of recurrence (except for skin basal-cell carcinoma and in-situ carcinoma including squamous cell carcinoma, bladder cancer in situ, endometrial cancer in situ, cervical cancer in situ/atypical hyperplasia, prostate cancer incidental finding (T1a or T1b), or breast cancer in situ) within 5 years prior to the first dose of study drug.
  12. Active GI dysfunction interfering with the ability to swallow tablets, or any GI dysfunction that could interfere with absorption of study treatment.
  13. Grade ≥ 3 peripheral neuropathy, and Grade ≥ 2 painful neuropathy, within 3 weeks prior to the first dose of study drug.
  14. Previous history of deep vein thrombosis.
  15. Serious, active psychiatric, or medical conditions which, in the opinion of the Investigator, could interfere with study treatment.
  16. Participation in an investigational anti-cancer clinical study within 3 weeks or 5 half-lives (T1/2) prior to the first dose of study drug.
  17. Received ASCT within 12 weeks prior to the first dose of study drug or previous allogeneic stem cell transplantation (no time limitation).
  18. Treatment with an approved or trial anticancer drug was given within 4 weeks prior to the first study.
  19. Known intolerance to or contraindication for glucocorticoid therapy.
  20. Prior exposure to a SINE compound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Assessed from the date of first dose of study treatment until the date that PD assessed up to 12months
  ORR in each arm: partial response (PR) + very good partial response (VGPR) + complete response (CR)

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) | 12 months
  To evaluate the minimal residual disease in CR and sCR patients
Overall Survival (OS) | 12 months
  The estimates of Kaplan-Meier
Progression-Free Survival (PFS) | 12 months
  Duration from start of study treatment to PD or death (regardless of cause), whichever comes first
Duration of Response (DOR) | 12 months
  Duration from the first observation of at least PR to time of disease progression, or deaths due to disease progression,whichever occurs first.
Clinical Benefit Rate (CBR) | 12 months
  Clinical Benefit Rate (CBR=ORR+Minor Response [MR])
Disease Control Rate (DCR) | 12 months
  Disease Control Rate (DCR=CBR+Stable Disease[SD; for a minimum of 12 weeks])
Number of Participants with Adverse Events | From first dose of study drug administration to end of treatment (up to 12 months)
  Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, M.D., Ph.D, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD results are used for publication,and can be shared with other investigators and sponsors
Supporting Information: Study Protocol
Time Frame: Study Protocol can be shared Starting 12 months after publication
Access Criteria: Study Protocol must not be shared with non-participants until after publication and must be authorized by the principal investigator and sponsors

REFERENCES:
- [Derived] Peng L, Shan T, Zhou X, Feng Z, Qiang W, Lu J, He H, Du J. Lowering the Selinexor Dose within the Pomalidomide and Dexamethasone Combination Regimen Elicits Fewer Side Effects While Comparable Efficacy Against Relapsed/Refractory Multiple Myeloma. Onco Targets Ther. 2025 Jun 6;18:695-703. doi: 10.2147/OTT.S516486. eCollection 2025. PMID 40496494